CLINICAL TRIAL: NCT00775411
Title: Safety and Efficacy of a New Therapy as Adjunctive Therapy to Anti-vascular Endothelial Growth Factor (Anti-VEGF) in Subjects With Wet Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206207-019
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Choroidal Neovascularization; Age-Related Maculopathy
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — Dexamethasone; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 700 µg dexamethasone and ranibizumab (Experimental): 700 µg dexamethasone intravitreal injection at Day 1 in the study eye. Ranibizumab injection at Week 2 or 3 per specified criteria and starting at Week 4 at the investigator's discretion in the study eye.
  Interventions: Drug: dexamethasone; Biological: ranibizumab

INTERVENTIONS:
Drug: dexamethasone — 700 µg dexamethasone intravitreal injection at Day 1 in the study eye.
  Other Names: Posurdex
Biological: ranibizumab — Ranibizumab injection at Week 2 or 3 per specified criteria and starting at Week 4 at the investigator's discretion in the study eye.
  Other Names: Lucentis®

SUMMARY:
The study will evaluate the safety and efficacy of the intravitreal dexamethasone implant as adjunctive therapy to Anti-VEGF treatment in the study eye of treatment naïve subjects with choroidal neovascularization secondary to age-related macular degeneration. Subjects will be followed for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older with active subfoveal choroidal neovascularization (CNV) secondary to AMD
* Central retinal thickness ≥ 300 µm
* Visual acuity between 20/400 and 20/32
* Eligible for Anti-VEGF therapy

Exclusion Criteria:

* Previous treatment for CNV due to AMD
* High eye pressure
* Glaucoma
* Uncontrolled systemic disease
* Known allergy to the study medications
* Recent eye surgery or injections in the eye
* Female subjects that are of childbearing potential

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (3):
- San Antonio, Texas, United States
- Sydney, New South Wales, Australia
- Manila, Philippines

RESULTS

PARTICIPANT FLOW:
Groups:
- 700 µg Dexamethasone + Ranibizumab: 700 µg dexamethasone intravitreal injection at Day 1 in the study eye. Ranibizumab injection at Week 2 or 3 per specified criteria and starting at Week 4 at the investigator's discretion.
Period: Overall Study
Arm/Group | 700 µg Dexamethasone + Ranibizumab
Started | 44
Completed | 43
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | 700 µg Dexamethasone + Ranibizumab
Number analyzed (Participants) | 44
Age Continuous [Mean (Standard Deviation); unit: Years] | 72.3 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Central Retinal Thickness as Measured by Optical Coherence Tomography (OCT) at Week 4
Description: Optical Coherence Tomography (OCT), a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina, was performed on the study eye after pupil dilation at baseline and Week 4.
Time Frame: Baseline, Week 4
Population: Participants from the Intent to treat Population consisting of all enrolled participants with data available at Week 4 for analyses.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | 700 µg Dexamethasone + Ranibizumab
Number analyzed (Participants) | 43
Microns
  Baseline | 360.9 (69.23)
  Change from baseline at Week 4 | -62.0 (78.68)

2. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) at Week 26
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Time Frame: Baseline, Week 26
Population: Intent to treat population consisting of all enrolled participants.
Measure: Mean (Standard Deviation); unit: Number of letters
Arm/Group | 700 µg Dexamethasone + Ranibizumab
Number analyzed (Participants) | 44
Number of letters
  Baseline | 46.5 (17.73)
  Change from baseline at Week 26 | 4.5 (9.62)

3. Secondary Outcome: Percentage of Participants With Fluorescein Leakage Improved, Unchanged and Worsened From Baseline as Assessed by Fluorescein Angiography at Week 26
Description: Fluorescein angiography (FA) is a technique for examining the circulation of the retina (and detecting any leakage) using a dye-tracing method. Photographs are taken with a specialized low-power microscope with an attached camera designed to photograph the interior of the eye, including the retina and optic disc. FA at Week 26 was compared to FA at Baseline. The percentage of participants in each of the following categories is reported: Improved (Leakage area decreased >=10%), Unchanged (Leakage area changed < 10%) and Worsened (Leakage area increased >=10%).
Time Frame: Baseline, Week 26
Population: Participants from the Intent to treat population consisting of all enrolled participants with data available for analysis at Week 26.
Measure: Number; unit: Percentage of participants
Arm/Group | 700 µg Dexamethasone + Ranibizumab
Number analyzed (Participants) | 43
Percentage of participants
  Improved | 74.4
  Unchanged | 18.6
  Worsened | 7.0

ADVERSE EVENTS:
Arm/Group | 700 µg Dexamethasone + Ranibizumab
Serious Adverse Events (participants affected / at risk) | 6/44
Other Adverse Events (participants affected / at risk) | 9/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 700 µg Dexamethasone + Ranibizumab (N=44)
Anaemia (Blood and lymphatic system disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Endophthalmitis (Infections and infestations) | 1 — Event not related to study drug or study procedure
Fall (Injury, poisoning and procedural complications) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 700 µg Dexamethasone + Ranibizumab (N=44)
Conjunctival haemorrhage (Eye disorders) | 6
Intraocular pressure increased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.